CLINICAL TRIAL: NCT00256334
Title: Resveratrol for Patients With Colon Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Chao Family Comprehensive Cancer Center, Cancer Center, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 05-20; 2005-4333 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Colon Cancer; Cancer
Keywords: Colon Cancer; Resveratrol; Clinical Trial; WnT signaling; Grapes; Cancer prevention
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resveratrol (Experimental): GM-CSF administration to all subjects in addition to chemotherapy treatment.
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — Patients were randomly assigned to one of four dose cohorts: plant-derived resveratrol tablets (purchased through the Life Extension Foundation, Scottsdale, AZ) at a dose of 80 mg/day, plant-derived resveratrol tablets at a dose of 20 mg/day, Grape Powder (GP) dissolved in water and taken orally (supplied by the California Table Grape Commission) at a dose of 120 g/day, and GP at a dose of 80 g/day.

SUMMARY:
Resveratrol is purported to possess cancer preventive activity, especially for colon cancer, though its mechanisms of action are not well defined. Resveratrol is found in the skin of grapes and has anti-oxidative and pro-apoptotic effects on cancer cell lines in vitro. The main dietary sources of resveratrol are grapes, grape products, and red wine, and small amounts may be found in mulberries. A prior report and compelling preliminary data from our laboratory suggest that resveratrol modulates Wnt signaling, a signaling pathway which is activated in over 85% of colon cancers. In this proposal, studies were performed to define the actions of resveratrol on the Wnt signaling pathway in a clinical trial in which patients with colon cancer received treatment with Resveratrol, and correlative laboratory studies examined its effects directly on colon cancer and normal colonic mucosa. These studies provided data on the mechanisms of resveratrol action and provided a foundation for future prevention trials, correlative studies and therapeutic clinical research with this agent.

DETAILED DESCRIPTION:
Patients will be treated with a two-week course of resveratrol. The initiation of the treatment will be approximately 14 days before standard of care surgical resection of tumor. Resveratrol will be ingested as 20 mg pills or in the form of freeze-dried grape extract which is prepared by the California Table Grape Commission used under GMP guidelines for human consumption.

The first two patients receiving resveratrol will be treated at a dose of 20 mg/day, the third and fourth patients at a dose of 80 mg/day, and the fifth and sixth patients with a dose of 160 mg/day. All patients receiving grape extract will receive 125 mg/day that will have to be mixed with one 8 oz glass of water. There will be no dose adjustments. If a patient has any side effects which are attributed to the resveratrol, it will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with colon cancer by colonoscopic biopsy and tissue obtained under UCI04-05.
* Patients with a plan for surgical resection at UCIMC within 2-4 weeks of enrollment.

Exclusion Criteria:

* Surgical resection to be performed at a facility other than UCIMC.
* Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that resveratrol modulates Wnt signaling in vivo in colon cancer and normal colonic mucosa | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall Holcombe, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

REFERENCES:
- [Result] Nguyen AV, Martinez M, Stamos MJ, Moyer MP, Planutis K, Hope C, Holcombe RF. Results of a phase I pilot clinical trial examining the effect of plant-derived resveratrol and grape powder on Wnt pathway target gene expression in colonic mucosa and colon cancer. Cancer Manag Res. 2009 Apr 3;1:25-37. PMID 21188121
- See also: Open Access article permitting unrestricted noncommercial use with proper citation. — http://www.dovepress.com/results-of-a-phase-i-pilot-clinical-trial-examining-the-effect-of-plan-peer-reviewed-article-CMR